CLINICAL TRIAL: NCT01919086
Title: Response Adapted Therapy With Bortezomib/Dexamethasone Followed by Addition of Lenalidomide in Non Responders as Initial Treatment for Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-064
Record Dates: First submitted 2013-08-07; First posted 2013-08-08 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma (MM)
Keywords: Bortezomib; Dexamethasone; Lenalidomide; 13-064
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Lenalidomide

ARMS (1):
- Patients with Multiple Myeloma (Experimental): This is a phase II, single center clinical trial designed to evaluate the response rate and toxicity of a response-adapted, sequential therapy, using bortezomib and dexamethasone, followed by the addition of lenalidomide in non-responders, in patients with untreated MM.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — Bortezomib SC (or IV if SC not tolerated) 1.5 mg/m^2, days 1, 8, 15 and 22
Drug: Dexamethasone — Dexamethasone 40 mg PO or IV days 1, 4, 8,15 and 22 or on a split-dose regimen. (20mg BIW).
Drug: Lenalidomide — Lenalidomide may be added to the patient's regimen at any time if there is evidence of hematologic disease progression

SUMMARY:
The purpose of this study is to see if researchers could get the same good results with less toxicity by using this new approach.

We already know that the three drugs bortezomib, lenalidomide, and dexamethasone given together at the same time are effective. Most physicians therefore treat patients with multiple myeloma with the 3 drug combination. However, the researchers also know that the three drugs given together result in more side effects than when only 2 drugs (bortezomib and dexamethasone or lenalidomide and dexamethasone) are given. The researchers believe that all patients may not necessarily need the three drugs to have good results. In this study, the researchers will first treat your disease with bortezomib and dexamethasone. If the disease is not well controlled with these 2 drugs, only then the third drug, lenalidomide, will be added. By using this sequential approach we may reach the same good results with fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or greater at the time of signing the informed consent document.

  • Patients diagnosed with symptomatic multiple myeloma based on IMWG Diagnostic Criteria. According to these criteria, patient must have
  * Monoclonal plasma cells in the bone marrow ≥ 10% and/or presence of a biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma defining events:
  * Clonal bone marrow plasma cell percentage ≥ 60% (Note: clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate, the highest value should be used)
  * Involved:Uninvolved serum free light chain ratio ≥ 100 (values are based on the serum Freelite assay) The involved free light chain must be ≥ 10 mg/dL >1 focal lesions on MRI studies (each focal lesion must be 5 mm or more in size)
  * [C] Calcium elevation in the blood, defined as serum calcium >11 mg/dl or > 1 mg/dL higher than the upper limit of normal
  * [R] Renal insufficiency, defined as serum creatinine > 2 mg/dl or creatinine clearance < 40 mL/min
  * [A] Anemia, defined as hemoglobin <10 g/dl or > 2 g/dl below the lower limit of normal
  * [B] Lytic bone lesions or osteoporosis. one or more osteolytic lesions on skeletal radiography, CT, or PET-CT (if bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement)
* Patients must have symptomatic multiple myeloma without advanced organ damage (such as multiple fractures or advanced bone disease causing immobilization, renal failure, spinal cord compression, or organ compromise due to soft tissue plasmacytoma). If immediate therapy with radiation and high-dose steroids (eg, for spinal cord compression) or if triple therapy is clearly advisable from the start, the patient is not eligible for this trial.
* Patients with measurable disease defined as one or more of the following: serum M protein ≥ 1.0 g/dl, urine M-protein ≥ 200 mg/24h, and/or serum FLC assay: involved FLC level ≥ 10 mg/dl with abnormal serum FLC ratio.
* Only non transplant candidates or those who opt to forgo ASCT during first line therapy are eligible
* ECOG performance status ≤ 2
* Female patients must:

  * be postmenopausal for at least 1 year before the Screening visit, OR
  * be surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study treatment, OR
  * Agree to completely abstain from heterosexual intercourse
* Patients must be able to provide voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Participant treated with any prior systemic therapy with the exception of the following:

  * Treatment by localized radiotherapy for a specific indication within 2 weeks of initiation of treatment.
  * Treatment with corticosteroids, not to exceed the equivalent of 160 mg of dexamethasone over a four-week period before initiation of protocol therapy.
* Presence of Primary or associated amyloidosis (AL)
* Participants who plan to proceed with ASCT as part of first line therapy
* Poor tolerability or known allergy to lenalidomide, bortezomib and/or dexamethasone or compounds that have similar chemical or biologic composition to these study drugs.
* Platelet count < 50,000/mm3 within 21 days of initiation of protocol therapy for patients in whom <50% of bone marrow nucleated cells are plasma cells; or platelet count <30,000/mm3 for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells. Transfusion is not allowed to meet platelet eligibility criteria.
* ANC < 1,000 cells/mm3 within 21 days of initiation of protocol therapy. Growth factor administration is not allowed to meet ANC eligibility criteria.
* Hemoglobin < 8 g/dL within 21 days of initiation of protocol therapy. Transfusion may be used to meet hemoglobin eligibility criteria.
* Hepatic impairment, defined as bilirubin > 1.5 x institutional upper limit of normal (ULN) Patients with benign hyperbilirubinemia (e.g., Gilbert's syndrome) are eligible or AST (SGOT), or ALT (SGPT), or alkaline phosphatase ≥ to 2 x ULN, within 21 days of initiation of protocol therapy.
* Renal insufficiency, defined as creatinine clearance < 30 ml/min within 21 days of initiation of protocol therapy. Creatinine clearance will be the primary eligibility criteria in determining renal insufficiency. The Cockcroft-Gault formula.
* Active hepatitis B or C infection
* HIV 1 or 2 positivity
* Female participant who is pregnant or breast-feeding.
* Inability to comply with an anti-thrombotic treatment regimen (e.g., administration of aspirin, enoxaparin, or low molecular weight heparin administration).
* Peripheral neuropathy ≥ Grade 2 on clinical examination, within 21 days of initiation of protocol therapy.
* Participant who had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Participant who has hypersensitivity to bortezomib, boron, or mannitol.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Participant diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy. Patients who have had prior malignancies within the past 2 years but are considered to be "cured" with a low likelihood of recurrence may be eligible at the discretion of the Principal Investigator.
* Any other medical condition or laboratory evaluation that, in the treating physician's or principle investigator's opinion, makes the patient unsuitable to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
overall response rate | 2 years
  (defined as > or = to PR) after 4 cycles of response-adapted sequential therapy, using bortezomib and dexamethasone (BD) followed by the addition of lenalidomide in suboptimal responders

SECONDARY OUTCOMES:
overall response rate | 2 years
  for the entire population after up to 8 cycles of response-adapted sequential therapy
response | 2 years
  will be tabulated after the completion of cycle four and cycle eight (for those who would have completed 8 cycles), and the overall response rate for the entire population after up to eight cycles will be estimated and compared to the responses reported in the phase II study by Richardson et al. using the 3-drug-combination.
toxicity | 2 years
  Before each drug dose, the patient will be evaluated for possible toxicities that may have occurred after the previous dose(s). Toxicities are to be assessed according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), Version 4.0.
quality of life (QOL) | 2 years
  QoL will be assessed in this study using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) and its corresponding multiple myeloma module (EORTC QLQ-MY20).
progression-free survival (PFS) | 2 years
  will be estimated for all patients using Kaplan-Meier methodology. This analysis will include all patients regardless of their transplantation status.
Characterization of genomic mutations of targetable genes | 2 years
Characterization of immunomodulatory checkpoint pathways in multiple myeloma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/